CLINICAL TRIAL: NCT00864903
Title: A Comparison Between a New Experimental Enzymatic Assay to Real Time PCR for the Diagnosing of Central Nervous System Enteroviral Infection
Brief Title: A New Enzymatic Assay for Rapid Diagnosing of Central Nervous System Enteroviral Infection
Status: Withdrawn | Type: Observational
Why Stopped: The enzymatic assay was not sensitive nor spesific for the test.
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Dr. Yechiel Schlesinger, MD / Head of Infectious Diseases Unit, Shaare Zedek Medical Center
Other Study IDs: SZMC
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2009-03

CONDITIONS: Viral Meningitis
Keywords: enterovirus; aseptic meningitis; real time PCR; diagnostics
MeSH Terms: conditions — Meningitis, Viral; Enterovirus Infections; Meningitis, Aseptic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal Fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pediatric ER: any child undergoing a spinal tap due to suspected meningitis

SUMMARY:
A new enzymatic assay was developed by NMD Diagnostics for rapid diagnosis of Enteroviral CNS infection. This study will compare this assay to RT-PCR, by testing human CSF samples taken from children at the ER who are undergoing a spinal tap due to suspicion of meningitis.

DETAILED DESCRIPTION:
MND's new enzymatic assay is based on the detection of a specific viral enzyme through the detection of its enzymatic reaction. The detection of a specific enzymatic reaction is indicative to the presence of the specific virus in a biological specimen. This study will compare this diagnostic assay to RT-PCR for diagnosis of enteroviral infection in cerebrospinal fluid. CSF samples will be taken from children undergoing a spinal tap at the pediatric ER due to a suspicion of meningitis. A total of 100 samples will be collected, from children 0-16 years old who's parents agreed on participation in the study. A comparison of the enzymatic assay to RT-PCR as well as calibration and validation of the new assay will be done with the harvested samples, for a rapid and accurate identification of Enterovirus in human cerebrospinal fluid.

ELIGIBILITY:
Inclusion Criteria:

* any child undergoing a spinal tap
* parents agreed on participation

Exclusion Criteria:

* refusal to participate in the study

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children age 0-16 years who undergo a spinal tap at the pediatric ER due to suspected meningitis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yechiel Schlesinger, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (2):
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem
  - MND Diagnostics, Ness Ziona